CLINICAL TRIAL: NCT05751096
Title: Low-Intensity Focused Ultrasound For Insular Neuromodulation in Chronic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carilion Clinic (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-22-1597
Record Dates: First submitted 2023-02-06; First posted 2023-03-02 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Fibromyalgia; Complex Regional Pain Syndromes; Chronic Pain
MeSH Terms: conditions — Fibromyalgia; Complex Regional Pain Syndromes; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Participants will act as their own control with a cross over study design. LIFU application vs Sham will be applied on separate study days for both pain cohorts (FM and CRPS).
Who Masked: Participant
Masking Description: LIFU vs SHAM application study visit will appear identical to study participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- LIFU - CRPS (Active Comparator): Real LIFU application for CRPS cohort.
  Interventions: Device: Low-intensity Focused Ultrasound (LIFU)
- SHAM - CRPS (Sham Comparator): Sham LIFU application for CRPS cohort.
  Interventions: Device: Sham Low-intensity focused ultrasound (LIFU)
- LIFU - FM (Active Comparator): Real LIFU application for FM cohort.
  Interventions: Device: Low-intensity Focused Ultrasound (LIFU)
- SHAM - FM (Sham Comparator): Sham LIFU application for FM cohort.
  Interventions: Device: Sham Low-intensity focused ultrasound (LIFU)

INTERVENTIONS:
Device: Low-intensity Focused Ultrasound (LIFU) — repeat pulse application of low intensity focused ultrasound using a single element transducer to a selected neurological target for neuromodulation.
  Arms: LIFU - CRPS; LIFU - FM
Device: Sham Low-intensity focused ultrasound (LIFU) — Sham application of LIFU.
  Arms: SHAM - CRPS; SHAM - FM

SUMMARY:
Study investigating the potential benefit for chronic pain patients (CRPS and FM) using low-intensity focused ultrasound for neuromodulation.

DETAILED DESCRIPTION:
Before coming up with a low-intensity focused ultrasound (LIFU) therapy for complex regional pain syndrome (CRPS) and fibromyalgia (FM) by running a clinical trial, the investigators must run a proof-of concept study to understand whether LIFU neuromodulation will elicit behavior and physiological responses in both these populations. The first study will be to run a counterbalanced within subject design, of active or inactive LIFU. The order of the sham vs real LIFU will be randomized on separate visits. The primary objective is to test if LIFU will reduce pain sensation and a secondary objective to test if LIFU will improve clinical outcomes, including changes in skin temperature and swelling circumference (in centimeters) of the target limb. The target limb is defined for CRPS as the injured extremity (upper or lower limb) and for FM as the dominant upper extremity. These clinical outcomes are common for both CRPS and FM population, along with pain, and these measurements are being taken to see if LIFU will affect these clinical features. LIFU has been tested extensively on healthy participants, demonstrating changes in brain activity without any damage.

An ultrasound transducer is the device used to apply LIFU, which will be fitted onto the scalp using a real-time head tracking infrared camera. Brief low-intensity ultrasound pulses will be delivered. Quantitative sensory testing (QST) will be utilized to cause a pain response by placing a thermode on the skin of the hand, forearm, lower leg, or foot and the temperature will be raised or lowered at a set rate. There will be four separate QST protocols including thermal thresholding, conditioned pain modulation (CPM), temporal summation of pain (TSP) and contact heat provoked potential (CHEP).

Thermal pain threshold testing will be established on the target limb to determine the individualized baselines for additional testing protocols. The QST device will be set to a baseline temperature of 32° C and increased at a rate of 1° C/sec. Once the participant feels pain from the heat stimulus, a button that returns the temperature to baseline will be pressed. This process will repeat 5 times and the average threshold will be calculated. CPM involves the co-delivery of a conditioned stimulus and a test stimulus. For the conditioned cold stimulus, the patients will submerge their opposite limb (of target limb) in a bucket of ice water, and it will be followed by the test stimulus, a heat stimulus to the target limb. The patients will then rate the perceived pain on a 10-point scale and the entire procedure will be repeated 3 times before and after LIFU stimulation. For TSP, heat stimulation is applied to the selected site. The baseline is set and is increased up to a destination temperature determined by individuals threshold testing and then either remains constant or pulses for up to 180 seconds. Subjects will rate the magnitude of perceived pain either verbally or numerically using a 10-point scale and the procedure will be performed 3 times before and after LIFU stimulation. For CHEP, the heat stimuli are given at random intervals between 10-20 seconds on multiple varied locations on the target limb to avoid habituation and heating. Patients will rate 40 stimuli on a perceived pain 10-point scale before and after LIFU stimulation and brain responses recorded using electroencephalography (EEG).

Non-contact infrared thermometers will be used to take skin temperature of the target limb and soft tape measures will be used to measure (in centimeters) the largest circumference (region of inflammation for CRPS patients and variable for FM patients depending on which muscle is larger) of the target limb.

A total of 15 CRPS patients and 12 FM patients will be enrolled in the study, with the Carilion Clinic Pain Management physicians using the established Budapest Criteria to diagnose CRPS type I and type II. The first session will involve obtaining MRI and CT anatomical scans, needed to accurately target the area of interest (anterior insula) during the QST sessions and ensure accurate application of the LIFU for each individual. Baseline clinical measurements of the target limb will also be obtained. The next two sessions will be randomly counterbalanced with LIFU or sham while obtaining QST and clinical measurements. Blood pressure, respiratory rate, galvanic skin response, photoplethysmography, and two-lead electrocardiogram will also be collected to monitor the patient's autonomic nervous system changes as potential confounding factors as well as assessing for effects from the ultrasound. Questionnaires will be administered via Redcap throughout each session to document potential confounding factors such as depression, fear and anxiety while also recording the patient's symptoms before and after LIFU application. Brief pain inventory (BPI) will also be documented for the CRPS participants, measuring both the intensity of pain and the interference of pain in the patient's life along with the revised fibromyalgia impact questionnaire (FIQR) for the FM participants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of complex regional pain syndrome (CRPS) I or II (Budapest Criteria) by Carilion physician. OR Diagnosis of fibromyalgia (FM) by Carilion physician (American College of Radiology 2011 modified fibromyalgia criteria).

Exclusion Criteria:

* Contraindications to MRI.
* Contraindications to CT
* History of seizures and/or pseudo-seizures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Perceived Pain scores | through study completion, an average of 2 weeks.
  Patients will rate their perceived pain (on a 0-9 scale, no pain - severe pain) before and after application of LIFU or Sham

SECONDARY OUTCOMES:
Clinical outcome - skin temperature | through study completion, an average of 2 weeks
  Skin temperature of affected limb will be measured (celsius)
Clinical outcomes - circumference | through study completion, an average of 2 weeks
  swelling circumference of affected limb will be measured (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Stringer, MD, Principal Investigator — Carilion Clinic
Locations (1):
- Fralin Biomedical Research Institute, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No